CLINICAL TRIAL: NCT04860505
Title: Combo-PEP: Multipurpose Prevention of Post-Exposure Prophylaxis Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen Kelley, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002242; 0000058968 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Sexually Transmitted Diseases
Keywords: Post-Exposure Prophylaxis; HIV; STI; PEP; Prevention
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Doxycycline; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doxycycline and Biktarvy (Experimental): Participants will take both study drugs simultaneously at home approximately 1 hour before Visit 2 and will be instructed to take a timestamped photograph or videotape of themselves taking the dose.
  Interventions: Drug: Doxycycline; Drug: Biktarvy

INTERVENTIONS:
Drug: Doxycycline — Doxycycline (DOX [200 mg]) is an oral medication used to treat or prevent infections that are strongly suspected to be caused by bacteria; it is an antimicrobial drug indicated for bacterial infections such as sexually transmitted infections.
Drug: Biktarvy — Biktarvy (200mg) is an oral combination anti-HIV medication that contains the drugs tenofovir alafenamide, emtricitabine, and bictegravir.

SUMMARY:
The study will determine tissue pharmacology of a single dose of doxycycline for sexually transmitted infection (STI) Post-exposure Prophylaxis (PEP).

DETAILED DESCRIPTION:
To determine tissue pharmacology of a single dose of doxycycline for STI PEP, investigators at Emory University will collaborate with the Centers for Disease Control and Prevention (CDC) to conduct a clinical trial of up to 20 men who have sex with men (MSM) and women aged 18-59, with measurement of anti-retroviral drug and doxycycline concentrations in the rectum and vaginal regions.

ELIGIBILITY:
Inclusion Criteria:

1. HIV negative person, who was assigned male or female at birth, who reports sex with another man in the last year and is in good general health
2. Aged 18-59 years
3. Not currently taking PrEP and no plans to initiate during study
4. Not currently taking PEP
5. Not currently taking doxycycline or other tetracycline-derived antibiotics and no plans to initiate during the study
6. Willing to use condoms consistently for the duration of the study
7. Able to provide informed consent in English
8. No plans for relocation in the next 4 months
9. Willing to undergo peripheral blood, urine, rectal or vaginal secretion collection, and a rectal or vaginal and cervical biopsy procedure
10. Willing to use study products as directed
11. Hepatitis B surface antigen (HBsAg) negative (screening lab test)
12. Creatinine clearance >60 ml/min

Exclusion Criteria:

1. Currently infected with hepatitis virus and/ or has liver disease
2. Current or chronic history of kidney disease or creatinine clearance (CrCl)<60 ml/min
3. Continued need for, or use during the 90 days prior to enrollment, of the following medications:

   1. Systemic immunomodulatory agents
   2. Supraphysiologic doses of steroids (short course steroids less than 7 days duration, allowable at the discretion of the investigators)
   3. Chemotherapy or radiation for treatment of malignancy
   4. Experimental medications, vaccines, or biologicals
4. Intent to use HIV antiretroviral pre/post-exposure prophylaxis (PrEP or PEP) during the study, outside of the study procedures
5. Intent to use doxycycline or other tetracycline-derived antibiotics during the course of the study, outside of the study procedures
6. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements
7. Not pregnant and no plans on getting pregnant throughout the duration of the study
8. Known allergic reaction to study drugs

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published for this study (including text, tables, figures, and appendices), will be made available for sharing, after de-identification.
Supporting Information: Study Protocol
Time Frame: Data will be made available to researchers providing a methodologically sound proposal, beginning 9 months and ending 36 months following publication.
Access Criteria: Proposals should be directed to colleen.kelley@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Hope Clinic in Atlanta, Georgia, USA. Participant enrollment began May 20, 2021 and all follow-up assessments were completed by May 9, 2022.
Groups:
- Doxycycline and Biktarvy: Participants took both study drugs simultaneously at home and came to the clinic for a study visit the following day for samples to be obtained 24 hours after the single dose of study drugs.
  Doxycycline (DOX [200 mg]) is an oral medication used to treat or prevent infections that are strongly suspected to be caused by bacteria; it is an antimicrobial drug indicated for bacterial infections such as sexually transmitted infections.
  Biktarvy (200mg) is an oral combination anti-HIV medication that contains the drugs tenofovir alafenamide, emtricitabine, and bictegravir.
Period: Overall Study
Arm/Group | Doxycycline and Biktarvy
Started | 20
Attended 24 Hours Post-dose Visit | 20
Completed (Completed 7 days post-dose visit) | 18
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Doxycycline and Biktarvy: Participants took both study drugs simultaneously at home and came to the clinic for a study visit the following day for samples to be obtained 24 hours after the single dose of study drugs.
Arm/Group | Doxycycline and Biktarvy
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Rectal Doxycycline Concentration
Description: Doxycycline concentration in tissue from a rectal biopsy was measured. Rectal biopsies were obtained from men. Women had the option to provide a rectal tissue sample.
Time Frame: 24 hours after a single dose
Population: This analysis includes participants who completed the rectal biopsy during the 24-hours post-dose visit. Ten men and 5 women provided rectal tissue samples at the 24-hours post-dose visit. One male attended the visit but was not able to tolerate the biopsy procedure and no rectal tissue was obtained.
Measure: Median (Full Range); unit: µg/g
Arm/Group | Doxycycline and Biktarvy
Number analyzed (Participants) | 15
µg/g | 0.654 [0.305 to 1.237]

2. Primary Outcome: Vaginal Doxycycline Concentration
Description: Doxycycline concentration in tissue from a vaginal biopsy was measured.
Time Frame: 24 hours after a single dose
Population: One female attended the visit 24 hours post-dose but was not able to proceed with the vaginal biopsy procedure due to menses and vaginal rugae.
Measure: Median (Full Range); unit: µg/g
Arm/Group | Doxycycline and Biktarvy
Number analyzed (Participants) | 8
µg/g | 0.367 [0.203 to 1.445]

3. Primary Outcome: Plasma Doxycycline Concentration
Description: Doxycycline concentration in plasma was measured.
Time Frame: 24 hours after a single dose
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Doxycycline and Biktarvy
Number analyzed (Participants) | 20
µg/mL | 487 [305 to 824]

4. Secondary Outcome: Rectal Bictegravir Concentration
Description: Bectegravir concentration in tissue from a rectal biopsy was measured.
Time Frame: 24 hours after a single dose
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/g
Arm/Group | Doxycycline and Biktarvy
Number analyzed (Participants) | 15
µg/g | 0.085 [NA to 0.391] — The lowest value is below the limit of detection of 0.010.

5. Secondary Outcome: Vaginal Bictegravir Concentration
Description: Bictegravir concentration in tissue from a vaginal biopsy was measured.
Time Frame: 24 hours after a single dose
Population: as for outcome 2
Measure: Median (Full Range); unit: µg/g
Arm/Group | Doxycycline and Biktarvy
Number analyzed (Participants) | 8
µg/g | 0.207 [NA to 1.038] — The lowest value is below the limit of detection of 0.010.

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of enrollment until the participants completed the study or withdrew from the study, up to 7 days.
Arm/Group | Doxycycline and Biktarvy
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT04860505/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT04860505/ICF_001.pdf